CLINICAL TRIAL: NCT02923141
Title: Trauma Intervention for Affect Regulation, AIDS, and Substances
Acronym: TIARAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Carrico, Associate Professor of Public Health Sciences and Psychology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20160744
Record Dates: First submitted 2016-09-28; First posted 2016-10-04 (Estimated); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Human Immunodeficiency Virus; Substance Related Disorder; Post Traumatic Stress Disorder
Keywords: substance use; trauma; HIV; viral load; women
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Substance-Related Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neutral Writing + Contingency Management (Active Comparator): Participants will attend four attention-matched control sessions, consisting of face-to-face administration of psychological measures and neutral writing exercises. Participants will also take part in 36 contingency management sessions in which they provide self-collected urine for toxicology screening and receive financial incentives for each negative drug result.
  Interventions: Behavioral: Neutral Writing; Behavioral: Contingency Management
- Expressive Writing + Contingency Management (Active Comparator): Participants will attend four expressive writing sessions focusing on traumatic or stressful events. Participants will also take part in 36 contingency management sessions in which they provide self-collected urine for toxicology screening and receive financial incentives for each negative drug result.
  Interventions: Behavioral: Expressive Writing; Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Neutral Writing
  Arms: Neutral Writing + Contingency Management
Behavioral: Expressive Writing
  Arms: Expressive Writing + Contingency Management
Behavioral: Contingency Management

SUMMARY:
The Purpose of this study is to see if it is possible to deliver an intervention that targets trauma, substance use, and engagement in HIV care with HIV-positive women.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* woman or trans woman
* substance use
* elevated PTSD symptoms
* HIV care difficulties

Exclusion Criteria:

* not HIV positive
* no substance use
* men
* no HIV care difficulties
* no history of trauma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as a woman (cisgender or transgender)
Enrollment: 16 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Reduction in HIV RNA Copies/mL | 6 months

SECONDARY OUTCOMES:
Increase in T-helper (CD4+) cell count | 6 months
Reduction in HIV transmission risk | 6 months
  self-reported condomless, serodiscordant sex and HIV viral load greater than 200 copies/mL
Decrease in stimulant use | 6 months
  self-report
Decrease in stimulant use | 6 months
  urine toxicology screening
Decrease in post-traumatic stress disorder (PTSD) symptoms | 6 months
  self-report measure: PTSD Checklist for DSM-5
Decrease in depressive symptoms | 6 months
  self-report measure: Centers for the Epidemiologic Study of Depression (CES-D)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Carrico, Ph.D., Principal Investigator — University of Miami
Locations (1):
- Clinical Research Building, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jemison D, Jackson S, Oni O, Cats-Baril D, Thomas-Smith S, Batchelder A, Rodriguez A, Dilworth SE, Metsch LR, Jones D, Feaster DJ, O'Cleirigh C, Ironson G, Carrico AW. Pilot Randomized Controlled Trial of a Syndemics Intervention with HIV-Positive, Cocaine-Using Women. AIDS Behav. 2019 Sep;23(9):2467-2476. doi: 10.1007/s10461-019-02625-2. PMID 31407212